CLINICAL TRIAL: NCT02159482
Title: Pilot Study of Interferon Alfa for Patients Who Have Received Cancer Vaccines
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low enrollment
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00014489
Record Dates: First submitted 2014-06-06; First posted 2014-06-10 (Estimated); Results first posted 2014-07-16 (Estimated); Last update posted 2014-07-25 (Estimated); Status verified 2014-06

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — Interferon alpha-2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- interferon-alfa-2a (Experimental): Starting within 6 months after completion of the dendritic cell vaccine, a dose of interferon alfa-2a will be administered subcutaneously in the skin of the arm, thigh or abdomen every other day for a total of 6 injections.
  Interventions: Drug: Interferon Alfa-2a

INTERVENTIONS:
Drug: Interferon Alfa-2a
  Other Names: Roferon®-A

SUMMARY:
This research study is for people who have previously received cancer vaccines. The investigators are testing a form of therapy known as interferon alfa-2a, which is commercially available as the drug Roferon®-A, to see if it can be used to help boost the effects of the cancer vaccine and help the immune system attack the cancer.

It is believed that the body's immune system can attack tumor cells and kill them. This is thought to be due to immune cells called T cells which can recognize special proteins on the surface of tumors as a signal to fight the cancer. However, the vaccine may not work very well if the protein signal is too weak for the T cells to find your tumors. The investigators think that interferon alfa-2a can signal the cancer cells in the body to make more proteins that may allow the T cells to recognize and kill the cancer cells better.

ELIGIBILITY:
Inclusion Criteria:

* Must have received a cancer vaccine targeting tumor antigen.
* 6 months following the last dose of the prior vaccine.
* Measurable disease defined by the RECIST criteria (lesions that can be accurately measured in at least one dimension with the longest diameter ≥ 20 mm using conventional techniques or ≥ 10 mm with spiral CT.)
* Karnofsky performance status greater than or equal to 70%
* Estimated life expectancy > 6 months.
* Age ≥ 18 years.
* Adequate, hematologic function with:

  * WBC ≥ 3000 mm3
  * hemoglobin ≥ 9 mg/dL (may transfuse or use erythropoietin to achieve this level)
  * platelets ≥ 100,000/mm3
* Adequate, renal and hepatic function with:

  * serum creatinine < 2.5 mg/dL
  * bilirubin < 2.0 mg/dL
  * SGOT/SGPT < 1.5 x upper limit of normal
* No prior grade 3 or 4 major organ or allergic toxicity attributable to the prior vaccine
* Ability to understand and provide signed informed consent that fulfills Institutional Review Board guidelines.
* Ability to return to Duke University Medical Center for adequate follow-up, as required by this protocol.

Exclusion Criteria:

* Patients with concurrent chemotherapy, radiation therapy, or immunotherapy should be excluded. Patients may not have received interferon previously.
* Patients with either previously irradiated or new CNS (central nervous system) metastases at entry are excluded. Pre-enrollment head CT is not required if not indicated by clinical signs or symptoms.
* Patients with a history of auto-immune disease, such as but not restricted to, inflammatory bowel disease, systemic lupus erythematosus, ankylosing spondylitis, scleroderma, or multiple sclerosis.
* Patients with serious intercurrent chronic or acute illness, such as cardiac disease, (NYHA class III or IV), hepatic disease, or other illness considered by the PI as unwarranted high risk for investigational drug treatment.
* Patients with a medical or psychological impediment to probable compliance with the protocol.
* Concurrent second malignancy other than non-melanoma skin cancer, or controlled superficial bladder cancer.
* Presence of an active acute or chronic infection including: an urinary tract infection, HIV (as determined by ELISA and confirmed by Western Blot) or viral hepatitis (as determined by HBsAg and Hepatitis C serology). HIV patients are excluded based on immuno-suppression, which may render them unable to respond to the vaccine; patients with chronic hepatitis are excluded because of concern that hepatitis could be exacerbated by the injections.
* Patients on steroid therapy (or other immuno-suppressives, such as azathioprine or cyclosporin A) are excluded on the basis of potential immune suppression. Patients must have had 6 weeks of discontinuation of any steroid therapy (except that used as pre-medication for chemotherapy or contrast-enhanced studies) prior to enrollment.
* Patients with egg allergies or allergies to any component of the vaccine should be excluded from the protocol.
* Pregnant and nursing women should be excluded from the protocol since this research may have unknown and harmful effects on an unborn child or on young children. If the patient is sexually active, the patient must agree to use a medically acceptable form of birth control in order to be in this study. It is not known whether the treatment used in this study could affect the sperm and could potentially harm a child that maybe fathered while on this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2005-11; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Morse, MD, Principal Investigator — Duke University

RESULTS

PARTICIPANT FLOW:
Groups:
- Interferon-alfa-2a: Starting within 6 months after completion of the dendritic cell vaccine, a dose of interferon alfa-2a will be administered subcutaneously in the skin of the arm, thigh or abdomen every other day for a total of 6 injections.
  Interferon Alfa-2a
Period: Overall Study
Arm/Group | Interferon-alfa-2a
Started | 11
Completed | 6
Not Completed | 5
Not completed — Withdrawal by Subject | 2
Not completed — Physician Decision | 3

BASELINE CHARACTERISTICS:
Arm/Group | Interferon-alfa-2a
Number analyzed (Participants) | 11
Age, Customized [Number; unit: participants]
  18 years and older | 11
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 9
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 11

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Clinical Responders (Complete Response + Partial Response)
Description: Response determination will be made according to the RECIST criteria. Complete response defined as the disappearance of target lesion, confirmed at 1-4 weeks. Partial response defined as 30% decrease in longest dimension of target lesion, confirmed at 1-4 weeks.
Time Frame: 4 weeks
Measure: Number; unit: percentage of participants
Arm/Group | Interferon-alfa-2a
Number analyzed (Participants) | 6
percentage of participants | 0

2. Secondary Outcome: Proportion of Patients Experiencing an Increase in the Magnitude of the Tumor Antigen-specific Immune Response
Description: The proportion of patients experiencing an increase in the magnitude of the tumor antigen-specific immune response following the administration of interferon will also be estimated. Immune response will be determined by ELISPOT analysis.
Time Frame: 4 weeks
Population: Five subjects analysed due to one subject not completing blood draws.
Measure: Number; unit: percentage of participants
Arm/Group | Interferon-alfa-2a
Number analyzed (Participants) | 5
percentage of participants | 60

ADVERSE EVENTS:
Time Frame: 2 months
Description: An adverse event is any adverse change from the study subject's baseline (pre-treatment) condition, including any clinical or laboratory test abnormality that occurs during the course of the proposed clinical study after treatment has started.
Arm/Group | Interferon-alfa-2a
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 5/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Interferon-alfa-2a (N=6)
Platelet count decreased (Investigations) | 1 (1)
Fever (General disorders) | 2 (3)
fatigue (General disorders) | 4 (4)
Chills (General disorders) | 1 (2)
Flu like symptoms (General disorders) | 2 (2) — A disorder characterized by a group of symptoms similar to those observed in patients with the flu. It includes fever, chills, body aches, malaise, loss of appetite and dry cough.
Tongue swelling (General disorders) | 1 (1)
Injection site reaction (General disorders) | 1 (1) — A disorder characterized by an intense adverse reaction (usually immunologic) developing at the site of an injection.
Dry Mouth (Gastrointestinal disorders) | 1 (1)
Depression (Psychiatric disorders) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
anorexia (Metabolism and nutrition disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
diarrhea (Gastrointestinal disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Low accrual was due to a drug manufacturing issue.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes